CLINICAL TRIAL: NCT06743958
Title: Prehabilitative Training in Children and Adolescents With Soft Tissue or Bone Sarcoma of the Lower Extremity - a Feasibility Study
Brief Title: Prehabilitation in Childhood Soft Tissue or Bone Sarcomas
Acronym: Prehab4Kids
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Dr. von Haunersches Children's Medical Hospital, University of Munich, Germany (Other)
Responsible Party: Principal Investigator, Sabine Kesting, Head of Pediatric Exercise Oncology Working Group, Technical University of Munich
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Prehab4Kids
Record Dates: First submitted 2024-11-25; First posted 2024-12-20 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2024-11

CONDITIONS: Soft Tissue Sarcoma of the Lower Extremity; Bone Tumor of the Lower Extremity; Childhood and Adolescent Cancer
Keywords: prehabilitation; bone tumor; soft tissue sarcoma; exercise intervention; childhood cancer; functional outcomes
MeSH Terms: conditions — Bone Neoplasms; Sarcoma; Neoplasms

STUDY DESIGN:
Intervention Model Description: Bicentric feasibility trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Specific strength and balance training during neoadjuvant chemotherapy
  Interventions: Other: Exercise intervention
- Control group (No Intervention)

INTERVENTIONS:
Other: Exercise intervention — Specific strength and balance training intervention during neoadjuvant chemotherapy, twice per week for 30 min, progression according to individual status
  Arms: Intervention group

SUMMARY:
This study aims to investigate the feasibility of a prehabilitative training intervention. The intervention includes specific strength and balance exercises during neoadjuvant chemotherapy with children and adolescents diagnosed with soft tissue or bone tumor in the lower extremity. This explorative approach of prehabilitation might help to reduce muscle and bone weakening and associated functional limitations during and after acute therapy. By designing this study like a controlled clinical trials, the investigators will also gather preliminary data on the intervention's potential effects in enhancing/on the pre-operative condition. The goal is to improve post-operative outcome and rehabilitation processes in children and adolescents diagnosed with soft tissue or bone sarcoma of the lower extremity.

DETAILED DESCRIPTION:
Soft tissue and bone sarcomas of the lower extremity pose significant challenges for affected individuals, often associated with considerable burden. Chemotherapy, load restrictions, and surgery frequently result in long-term physical limitations, causing structural and functional deterioration. In childhood and adolescence, these challenges are particularly pronounced, as they affect physiological development, resilience, and autonomy. Although movement promotion and therapeutic programs are designed to address these deficits, they are typically implemented post-operatively and during follow-up care. The benefit of implementing a specific program before the operative therapy remains elusive. The presented study explores the feasibility of a supervised prehabilitative training intervention and gather preliminary data on its potential effects in enhancing the pre-operative condition. The goal is to improve post-operative outcome and rehabilitation in children and adolescents diagnosed with soft tissue or bone sarcoma of the lower extremity.

This bicentric feasibility study, designed as a controlled clinical trial, enrolls all children and adolescents aged 6-18 years who are newly diagnosed with primary osteosarcoma, Ewing's sarcoma, or rhabdomyosarcoma of the lower extremity. Based on the study site, participants are allocated to either the intervention group (IG) or control group (CG), with a target sample size of 16-18. The intervention consists of specific strength and balance training sessions during neoadjuvant therapy, conducted at least twice a week for a minimum of 30 minutes per session. The CG does not receive any training intervention. The study has been consented by the local ethics committee.

The primary endpoint is the proof of feasibility of the intervention, assessed via descriptive analysis of recruitment rate, acceptance, data quality, practicability, and safety (adverse events). The secondary endpoint is the demonstration of the efficacy of the intervention comparing structural and functional measurements intra-individually and between groups at four timepoints: within ten days post-diagnosis, pre-operatively (post-intervention), at the end of therapy, and at 1-year follow-up. The measurements include psoas muscle area, body composition, strength, mobility, balance ability, gait analysis, two questionnaires on physical activity and quality of life, and quantitative measures of the clinical course during treatment (days of hospitalization, infection rates, etc.).

This study is designed to evaluate the feasibility of a specific prehabilitative training intervention in children and adolescents with soft tissue or bone sarcoma of the lower extremity. Additionally, preliminary data on the effects of this training are collected, aiming to mitigate muscle mass loss, support physiological body composition, and improve functional outcomes such as balance, gait, and physical activity. Enhancing everyday functionality and fostering a sense of autonomy can significantly improve the quality of life in this population, underscoring the importance of investigating and promoting such interventions in this underrepresented patient group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a bone tumor or soft tissue sarcoma of the lower extremity
* Diagnosed less than 10 days ago, confirmed through biopsy
* Age Range of 6 to 18 years
* Treatment will be conducted at one of the two designated study sites

Exclusion Criteria:

* Medical contraindications for the implementation of the intervention and measurements, in consultation with the treating physicians (e.g., acute risk of bleeding or fractures, pain, infection, nausea, dizziness, lack of orthopedic clearance for weight-bearing in the tumor region, other acute orthopedic limitations unrelated to the underlying condition, etc.)
* Language barriers that prevent understanding of the instructions for study participation
* Cognitive impairment or developmental delay that hinders comprehension of the instructions in the testing situation, thereby preventing standardized diagnostic data collection and intervention

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility Criteria 1 - Recruitment Rate | At enrollment
  The number of children and adolescents diagnosed with bone and soft tissue sarcoma of the lower extremity who agree to participate compared to the total number approached for this study.
Feasibility Criteria 2 - Acceptance | From enrollment to 12 months following end of therapy
  Number of performed exercise sessions during intervention period compared to intended sessions and number of performed measurements and compared to intended measurements.
Feasibility Criteria 3 - Data Quality | From enrollment to 12 months following end of therapy
  Number of evaluable exercise documentation data and measurement data.
Feasibility Criteria 4 - Practicability | From enrollment to 12 months following end of therapy
  Difference between scheduled and required time frame for the exercise sessions and measurements.
Feasibility Criteria 5 - Participants' Feedback | From enrollment to 12 months following end of therapy
  Feedback questionnaire with multiple choice options and free text answers.

SECONDARY OUTCOMES:
Total psoas muscle area | From enrollment to 12 months following end of therapy
  Total psoas muscle area at lumbal level (L4) analyzed via MRI or PET CT
Fat-free mass | From enrollment to 12 months following end of therapy
  The weight of all body components excluding fat, measured in kilograms, using bioimpedance analysis. Outcome measures 7.-11. will be combined to report body composition.
Fat mass | From enrollment to 12 months after end of therapy
  Total body fat weight, measured in kilograms, assessed via bioimpedance analysis. Outcome measures 7.-11. will be combined to report body composition.
Total body water | From enrollment to 12 months after end of therapy
  The proportion of total body water in kg, expressed as percentage, measured through bioimpedance analysis. Outcome measures 7.-11. will be combined to report body composition.
Body cell mass | From enrollment to 12 months after end of therapy
  The mass of metabolically active cells in the body, measured in kilograms, via bioimpedance analysis. Outcome measures 7.-11. will be combined to report body composition.
Phase angle | From enrollment to 12 months after end of therapy
  An indicator of cellular health and membrane integrity, measured in degrees using bioimpedance analysis. Outcome measures 7.-11. will be combined to report body composition.
Muscle strength | From enrollment to 12 months following end of therapy.
  Overall muscle strength measured by hand-grip dynamometry measured in kilograms. Reference values enable comparison with healthy children and adolescents. Higher scores imply increased muscle strength.
Range of motion of the adjacent joints | From enrollment to 12 months following end of therapy
  Range of motion of the adjacent joints measured with an analog goniometer in degrees. Higher numbers of degrees imply better range of motion.
Gait analysis | From enrollment to 12 months following end of therapy
  Gait analysis measured with a force plate to analyze how pressure is distributed during stance phases of walking (vertical ground reaction force during loading response, mid stance, terminal stance, toe off).
Path length | From enrollment to 12 months after end of therapy
  The total distance traveled by the center of pressure during balance assessment, measured in centimeters using a force plate. Outcome measures 15.-18. will be combined to report balance ability.
Mean velocity | From enrollment to 12 months after end of therapy
  The average speed of center of pressure shifts during balance assessment, measured in meters per second with a force plate. Outcome measures 15.-18. will be combined to report balance ability.
Sway angle | From enrollment to 12 months after end of therapy
  The angular deviation of the center of pressure from a neutral position during balance tasks, measured in degrees using a force plate. Outcome measures 15.-18. will be combined to report balance ability.
Equlibrium score | From enrollment to 12 months after end of therapy
  Calculated from the anterior-posterior and medial-lateral projection of the 90% Standard Ellipse and estimated height of center of gravity during balance tasks in percentage using a force plate. Outcome measures 15.-18. will be combined to report balance ability.
Level of physical activity | From enrollment to 12 months following end of therapy
  Level of physical activity before, during and following therapy measured with the standardized ActiOn questionnaire. This tool reports individual physical activity levels and enables evaluation of meeting physical activity recommendations for children and adolescents.
Quality of life | From enrollment to 12 months following end of therapy
  Quality of life during and following therapy measured with the standardized and validated KINDL questionnaire. This tool enables evaluation of quality of life compared to reference values of healthy children and adolescents. Higher scores imply higher self-reported quality of life.
Quantitative measures of clinical course during treatment | From enrollment to 12 months following end of therapy
  Quantitative measures of clinical course during treatment (days of hospitalization, infection rates, days between surgery and start of adjuvant chemotherapy, units of physiotherapy) documented via analog and digital clinical record. This information is individual and not comparable to any reference values, however, provides important information regarding medical treatment and recovery process.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Technical University of Munich, Germany; TUM School of Medicine and Health, Department of Pediatrics. German Center for Child and Adolescent Health (DZKJ), partner site Munich, Munich, Bavaria
  - Dr. von Haunersches Kinderspital, Munich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Winter CC, Muller C, Hardes J, Gosheger G, Boos J, Rosenbaum D. The effect of individualized exercise interventions during treatment in pediatric patients with a malignant bone tumor. Support Care Cancer. 2013 Jun;21(6):1629-36. doi: 10.1007/s00520-012-1707-1. Epub 2013 Jan 5. PMID 23292667
- [Background] Runco DV, Zimmers TA, Bonetto A. The urgent need to improve childhood cancer cachexia. Trends Cancer. 2022 Dec;8(12):976-979. doi: 10.1016/j.trecan.2022.07.005. Epub 2022 Aug 3. PMID 35931609
- [Background] Pilz F, Vill K, Rawer R, Bonfert M, Tacke M, Heussinger N, Muller-Felber W, Blaschek A. Mechanography in children: pediatric references in postural control. J Musculoskelet Neuronal Interact. 2022 Dec 1;22(4):431-454. PMID 36458382
- [Background] Lurz E, Patel H, Lebovic G, Quammie C, Woolfson JP, Perez M, Ricciuto A, Wales PW, Kamath BM, Chavhan GB, Juni P, Ng VL. Paediatric reference values for total psoas muscle area. J Cachexia Sarcopenia Muscle. 2020 Apr;11(2):405-414. doi: 10.1002/jcsm.12514. Epub 2020 Jan 9. PMID 31920002
- [Background] Gotte M, Gauss G, Dirksen U, Driever PH, Basu O, Baumann FT, Wiskemann J, Boos J, Kesting SV. Multidisciplinary Network ActiveOncoKids guidelines for providing movement and exercise in pediatric oncology: Consensus-based recommendations. Pediatr Blood Cancer. 2022 Nov;69(11):e29953. doi: 10.1002/pbc.29953. Epub 2022 Sep 8. PMID 36073842
- [Background] Gauss G, Beller R, Boos J, Daggelmann J, Stalf H, Wiskemann J, Gotte M. Adverse Events During Supervised Exercise Interventions in Pediatric Oncology-A Nationwide Survey. Front Pediatr. 2021 Aug 19;9:682496. doi: 10.3389/fped.2021.682496. eCollection 2021. PMID 34490156
- [Background] Garcia MB, Ness KK, Schadler KL. Exercise and Physical Activity in Patients with Osteosarcoma and Survivors. Adv Exp Med Biol. 2020;1257:193-207. doi: 10.1007/978-3-030-43032-0_16. PMID 32483741
- [Background] Furtado S, Errington L, Godfrey A, Rochester L, Gerrand C. Objective clinical measurement of physical functioning after treatment for lower extremity sarcoma - A systematic review. Eur J Surg Oncol. 2017 Jun;43(6):968-993. doi: 10.1016/j.ejso.2016.10.002. Epub 2016 Oct 14. PMID 27836415
- [Background] Ehrhardt MJ, Leerink JM, Mulder RL, Mavinkurve-Groothuis A, Kok W, Nohria A, Nathan PC, Merkx R, de Baat E, Asogwa OA, Skinner R, Wallace H, Lieke Feijen EAM, de Ville de Goyet M, Prasad M, Bardi E, Pavasovic V, van der Pal H, Fresneau B, Demoor-Goldschmidt C, Hennewig U, Steinberger J, Plummer C, Chen MH, Teske AJ, Haddy N, van Dalen EC, Constine LS, Chow EJ, Levitt G, Hudson MM, Kremer LCM, Armenian SH. Systematic review and updated recommendations for cardiomyopathy surveillance for survivors of childhood, adolescent, and young adult cancer from the International Late Effects of Childhood Cancer Guideline Harmonization Group. Lancet Oncol. 2023 Mar;24(3):e108-e120. doi: 10.1016/S1470-2045(23)00012-8. Epub 2023 Feb 14. PMID 37052966
- [Background] Bhagat A, Kleinerman ES. Anthracycline-Induced Cardiotoxicity: Causes, Mechanisms, and Prevention. Adv Exp Med Biol. 2020;1257:181-192. doi: 10.1007/978-3-030-43032-0_15. PMID 32483740
- [Background] Basteck S, Guder WK, Dirksen U, Krombholz A, Streitburger A, Reinhardt D, Gotte M. Effects of an Exercise Intervention on Gait Function in Young Survivors of Osteosarcoma with Megaendoprosthesis of the Lower Extremity-Results from the Pilot Randomized Controlled Trial proGAIT. Curr Oncol. 2022 Oct 14;29(10):7754-7767. doi: 10.3390/curroncol29100613. PMID 36290890